CLINICAL TRIAL: NCT04913493
Title: Use of Sublingual Microcirculation and FloTrac Monitoring During Major Vascular Surgery and Its Effect on Hospital Length of Stay: a Prospective Cohort Study
Brief Title: Use of Sublingual Microcirculation and FloTrac Monitoring During Major Vascular Surgery and Its Effect on Hospital LOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patient recruited
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLOMIC
Record Dates: First submitted 2021-04-27; First posted 2021-06-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2023-04

CONDITIONS: Carotid Artery Plaque; Aortic Aneurysm; Aneurysm
MeSH Terms: conditions — Carotid Stenosis; Aortic Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Patients will only receive FloTrac/Vigileo monitoring which is standard of care.
- Experimental group (Experimental): Patients will receive an additional medical imaging intervention. Namely sublingual microcirculation imaging with Cytocam-IDF.
  Interventions: Procedure: Cytocam-IDF

INTERVENTIONS:
Procedure: Cytocam-IDF — Patients receive an extra medical imaging test perioperatively with the Cytocam-IDF
  Arms: Experimental group

SUMMARY:
the aim of this study is to determine whether an intraoperative optimization protocol using the enhanced flow-based hemodynamic parameters of the FloTrac/Vigileo device in combination with intraoperative measurement of the sublingual microcirculation with the Cytocam-IDF device would result in an improvement in outcome in high-risk patients undergoing major vascular surgery, measured by the hospital LOS in comparison with intraoperative FloTrac/Vigileo monitoring alone.

The FloTrac/Vigileo device only needs standard arterial access for enhanced, flow-based hemodynamic monitoring. It is reported to be easy to use and easy to set up and calculates the stroke volume (SV) on the basis of the arterial waveform in combination with demographic data. Cardiac index (CI), stroke volume index (SVI) as an indicator for fluid status and stroke volume variation (SVV) as an indicator for fluid responsiveness during mechanical ventilation and sinus rhythm will be continuously measured during major vascular procedures, including carotid endarterectomy (CEA), open abdominal aortic aneurysm (AAA) repair , endovascular aneurysm repair (EVAR), thoracic endovascular aneurysm repair (TEVAR) and fenestrated endovascular aneurysm repair (FEVAR).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Males and females
* ASA III classification
* Written informed consent obtained by the patient
* Elective hospital admission for major vascular surgery procedures (CEA, open AAA, EVAR, TEVAR, FEVAR)

Exclusion Criteria:

* Age < 18 years
* Presence of permanent cardiac arrythmias
* Weight < 55kg and > 140kg
* Pregnancy
* Emergency surgery
* Minor vascular procedures
* Refusal or inability to provide written informed consent (language barrier, mental retardation, dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Number of hospitalisation days. (LOS) | up to 30 Days
  How long is the hospital Length-Of-Stay?

CONTACTS AND LOCATIONS:
Overall Officials: Hélène De Cuyper, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
Patients individual data will not be shared. Findings of the study will be published in a scientific article.